CLINICAL TRIAL: NCT06897618
Title: Effect of Culturally Tailored Diabetes Education on Self-Management Behaviors of Adult Hispanic Males With Type 2 Diabetes Mellitus
Brief Title: Culturally Tailored Diabetes Education on Self-Management of Adult Hispanic Males With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment challenges
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2025-0124
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus; Diabete Type 2
Keywords: Type 2 diabetes; Self-Management Behaviors; Culturally Tailored Diabetes Education
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Culturally Tailored Diabetes Education (Experimental): Five weeks of culturally tailored diabetes self-management education modeled after Association of Diabetes Care and Education Seven-item Framework (ADCES7).
  Interventions: Behavioral: Culturally tailored diabetes self-management education

INTERVENTIONS:
Behavioral: Culturally tailored diabetes self-management education — Five weeks of culturally tailored diabetes self-management education modeled after Association of Diabetes Care and Education Seven-item Framework (ADCES7).

SUMMARY:
Diabetes mellitus (DM) is a global public health concern. In the United States, adult Hispanic males are particularly vulnerable to type 2 diabetes mellitus and are more likely to develop complications and subsequently die from it, compared to non-Hispanic White males. Evidence suggests good self-management behaviors can potentially prevent disease-related complications and improve clinical outcomes. The American Diabetes Association and Association of Diabetes Care and Education Specialists have endorsed diabetes self-management education as a necessary component of care for all individuals living with the disease. However, adult Hispanic males with type 2 diabetes mellitus living in the Middle Atlantic Region of the U.S., especially those who are underserved, typically lack access to formal diabetes self-management education (DSME). Further, the majority have never participated in such educational activities. A large body of evidence suggests DSME can effectively improve self-management behaviors in diverse populations around the globe. The purpose of the proposed study is to examine the effect of culturally tailored diabetes education on self-management behaviors of adult Hispanic males, aged 18-64 years, with type 2 diabetes mellitus living in the Middle Atlantic Region of the U.S. This study can shed more light on the effectiveness of community-based, culturally tailored diabetes educational activities in this vulnerable population and guide future efforts towards enhancing self-management.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adult Hispanic males 18-64 at time of study intervention.
* Diagnosis Codes: Patients with self-reported diagnosis of T2DM without complex, co-morbid conditions such as severe kidney disease and terminal illnesses such as cancer.
* English or Spanish speaking

Exclusion Criteria:

* Outside the age range listed above
* Without a diagnosis of type 2 diabetes

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Adult Hispanic males 18-64 at time of study intervention
Enrollment: 40 (Actual)
Dates: Start 2025-09-12 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Healthy Eating | At baseline and right after the 5 week educational intervention
  Healthy eating behaviors will be measured by self-reported data on diet adherence utilizing scoring derived from the Spanish version of the Summary of Diabetes Self-Care Assessment (SDSCA) scale. Items 1-5 relate to dietary behaviors, for example, "how many of the last seven days have you followed a healthful eating plan?" Diet will be scored using the mean number of days for items 1-5, using a reverse score for item 4. Scores range from 0 to 7 with higher numbers corresponding to higher levels of self-care activity performance
Staying Active | At baseline and right after the 5 week educational intervention
  Physical activity behaviors will be measured by self-reported data on exercise adherence utilizing scoring derived from the Spanish version of the Summary of Diabetes Self-Care Assessment (SDSCA) scale. Items 6-7 pertain to exercise activity, for example, "on how many of the last seven days did you participate in at least 30 minutes of physical activity?" Exercise will be scored using the mean number of days for items 6 and 7. Scores range from 0 to 7 with higher numbers corresponding to higher levels of self-care activity performance
Medication Use | At baseline and right after the 5 week educational intervention
  Medication use behaviors will be measured by self-reported data on medication adherence utilizing scoring derived from the Spanish version of the Summary of Diabetes Self-Care Assessment (SDSCA) scale. Medication use will be scored using total number of days for item 12. Scores range from 0 to 7 with higher numbers corresponding to higher levels of self-care activity performance

CONTACTS AND LOCATIONS:
Overall Officials: Beryl O'Donnell, MSN, RN, NP-C, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack Meridian Health, JFK University Medical, Plainfield, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No